CLINICAL TRIAL: NCT06129773
Title: Comparison Of Outcome Of Antibiotic Coated Vicryl Vs Non-Coated Vicryl In Abdominal Fascial Closure After Laparotomy In Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Adeel Ashiq (Other)
Responsible Party: Sponsor-Investigator, Muhammad Adeel Ashiq, Dr Muhammad Adeel Ashiq, Children Hospital and Institute of Child Health, Lahore
Organization: Children Hospital and Institute of Child Health, Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Adeel1
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Surgical Site Infection
Keywords: SSIs, anti biotic coated vicryl, laparotomy, Triclosan coated vicryl, Vicryl plus, Surgical site infection, Uncoated vicryl,
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- anti biotic coated group (Experimental)
  Interventions: Procedure: antibiotic coated vicryl used for fascial closure
- non coated group (No Intervention)

INTERVENTIONS:
Procedure: antibiotic coated vicryl used for fascial closure — in this group fascial closure was done with antibiotic coated vicryl to compare with non coated vicryl after lapaprotomy in contaminated wounds
  Arms: anti biotic coated group

SUMMARY:
We are investigating outcome of antibiotic coated vicryl versus non coated vicryl in terms of rate of surgical site infection and lebgth of hospital stay in children after lalaprotomy for perforated viscera. total 100 patients will be taken and 50 in each group.

DETAILED DESCRIPTION:
Pneumoperitoneum is typically a surgical emergency, particularly in children and more than 90% of occurrences are caused by perforation of the gastrointestinal tract and other hollow viscera. Wound infections after abdominal surgery are still frequent types of nosocomial infections. Sutures can be a source of wound infection and dehisence due to bacterial adherence and colonization. Sutures coated with antibacterial agents have been developed in an attempt to reduce bacterial adherence and colonization of suture materials. The objective of the study is to compare the outcome of antibiotic coated vicryl versus non-coated vicryl in abdominal fascial closure after laparotomy in children in regards of surgical site infections. It will be a randomized controlled trial in which 100 patients admitted in Children Hospital Lahore will be included. Simple random sampling will be carried out. Informed written consent will be taken from patients' guardian. The patients will be divided into two groups (50 in each group). Group-A patients will undergo laparotomy closure with antibiotic coated vicryl while Group-B patient will experience non-coated vicryl in abdominal fascial closure. All patients will be examined on 3rd, 7th and 30th post-operative day for wound infection according to Southampton wound scoring system. Data will be collected through predesigned proforma, which will be entered and statistically analyzed using SPSS version 24.0. For quantitative variables mean and standard deviation will be calculated and for qualitative variables frequency and percentages will be calculated. Data will be presented in tables and graphs. Chi-square test will be used to estimate the association between qualitative variables. P-value <0.05 will be considered significant. It is expected that results of this study may be helpful for healthcare providers to provide appropriate treatment to the patients and to prevent them from wound related complications.

ELIGIBILITY:
Inclusion Criteria:

* • Children with pneumoperitoneum / perforated viscus

  * Children aged 0 day to 15 years
  * Both genders

Exclusion Criteria:

* • Malnourished children

  * Children aged above 15 years
  * Clean surgeries
  * Low Hb level
  * Parents unwilling to take part

Ages: 4 Hours to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Rate of surgical site infection | 30 days
  rate of surgical site infection will be measured in percentage

CONTACTS AND LOCATIONS:
Locations (1):
- The Children Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No